CLINICAL TRIAL: NCT07132203
Title: A Multicenter Trial for the Safety and Efficacy of a Magnetic Resonance-Guided Laser Interstitial Thermal Therapy for Brain Metastases
Brief Title: Magnetic Resonance-Guided Laser Interstitial Thermal Therapy for Brain Metastases Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Sinovation (Beijing) Medical Technology (Unknown)
Responsible Party: Principal Investigator, Wang Jia, Professor of Beijing Tiantan Hospital, Capital Medical University, Beijing Tiantan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QX2021-025-02
Record Dates: First submitted 2025-08-10; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Brain Metastasases
Keywords: laser interstitial thermal therapy; brain metastasases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- laser interstitial thermal therapy (Experimental): The subjects will undergo laser interstitial thermotherapy after the screening process is completed. There will be no restrictions on other treatment methods.
  Interventions: Device: Laser interstitial thermal therapy

INTERVENTIONS:
Device: Laser interstitial thermal therapy — The LITT procedure was performed using the LS1 laser ablation system and SR1 stereotactic robotic system (Sinovation, Beijing, China). The ablation system was equipped with a 980-nm laser with a maximum of 15 W of power, a core silica fiber optic with a 1.8-mm diameter cooling catheter, and a cooling pump to make saline flow into and out through the catheter. The optic and catheter approaches were planned with the preoperative simulation software (Sinovation, Beijing, China) using the preoperative T1-weighted MRI scan, and passing through important cerebral vascular and functional zones was avoided。. The catheter was implanted by neurosurgeons under stereotactic guidance, and a laser probe was inserted through the catheter. After LITT, a T1-weighted intraoperative MRI scan was performed to confirm the effect of ablation. The ablation rate was calculated by another neurosurgeon who did not participate in the study.

SUMMARY:
In accordance with the requirements of the "Good Clinical Practice for Medical Devices", this clinical trial is conducted to further evaluate the safety and efficacy of the magnetic resonance-guided laser ablation treatment system and the laser ablation minimally invasive treatment kit produced by Sinovation (Beijing) Medical Technology. This clinical trial adopts a multi-center, single-groupdesign. After all subjects sign the informed consent form and pass the screening, they will receive the implantation and treatment of the trial products. Follow-up visits will be conducted on the 2±1 day after the surgery, and the efficacy rate of ablation as assessed after the surgery was used as the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and above;
2. Previously diagnosed or newly diagnosed with a malignant tumor in the body accompanied by intracranial metastasis;
3. The lesion can be clearly identified in the magnetic resonance imaging, and the number of lesions does not exceed 4;
4. The lesion to be treated by ablation has a short axis of ≤ 30mm;
5. Karnofsky Performance Status (KPS) score ≥ 60;
6. The subject or their guardian can understand the purpose of the trial, demonstrate sufficient compliance with the trial protocol, and sign the informed consent form.

Exclusion Criteria:

1. Patients with contraindications for MRI;
2. Patients with severe coagulation dysfunction;
3. Pregnant or lactating women, and those planning to conceive within 6 months;
4. Patients with the longest axis of the maximum brain metastasis lesion less than 5mm;
5. Subjects who have participated in any clinical trials of drugs or medical devices within 3 months before screening;
6. Patients judged by the researcher to be unable to tolerate ablation treatment;
7. Patients judged by the researcher to have evidence of severe or uncontrollable systemic diseases;
8. Subjects considered by the researcher to be unsuitable for this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
The efficacy rate of ablation | within 2days post LITT
  The ablation results were evaluated by an independent third-party imaging review panel. Two junior physicians from the third-party review panel drew the boundaries of the brain metastases and the actual ablation areas separately, and when ≥ 90% of the tumor tissue was ablated, it was considered a complete surgical resection or near-complete resection, and the ablation was deemed effective.

SECONDARY OUTCOMES:
The rate of local control of the treated lesion | The 30th day after the operation, the 90th day after the operation, and the 180th day after the operation
  The RANO-BM standard was used for evaluation. Taking the MRI images of the lesion as the baseline, MRI images were re-scanned at 30 ± 7 days, 90 ± 7 days, and 180 ± 14 days after the operation. The total long diameter of the brain metastases before ablation and the total long diameter of the remaining lesions at each follow-up point after the operation were measured respectively. If the long diameter of the lesion could not be measured due to reasons such as lesion size, it was recorded as "unable to measure", and the assessment would be conducted again at the next follow-up. Taking the total long diameter of the brain metastases before ablation as the baseline, the total long diameter changes of the affected lesions were calculated, and finally, it was evaluated whether the affected lesions had progressed.
the progression free survival | up to 6 months
  The assessment of PFS is conducted using the standard RANO-BM criteria commonly used in neurosurgery. A comprehensive evaluation is carried out from the perspectives of target lesions, non-target lesions, new lesions, hormone use, and clinical symptoms to determine whether the patient's condition has progressed.
The overall survival | up to 6 months
  defined as the time period from the date of surgery to the death of the subject.
Karnofsky performance scale | The 30th day after the operation, the 90th day after the operation, and the 180th day after the operation
  The Karnofsky score runs from 100 to 0, where 100 is "perfect" health and 0 is death. Although practitioners occasionally assign performance scores in between standard intervals of 10.
The incidence of short-term complications | the day of operation and 2 days post poeration
  The expected possible complications include intracranial hemorrhage, infection, high fever, hemiplegia, intracranial edema, cerebrospinal fluid leakage, poor incision healing, epilepsy, memory loss, visual field loss, aphasia, mental disorder, coma; as well as secondary brain edema caused by thermal injury and the risk of corresponding inflammatory factor release
Adverse Event rate | up to 6 months
  Adverse Event refers to any adverse medical occurrence that occurs during a clinical trial, regardless of whether it is related to the device.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Jia, Principal Investigator — Beijing Tiantan Hospital
Locations (6):
- China (6):
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Jilin University-China-Japan Friendship Hospital, Changchun, Jilin
  - Huashan Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No
The test data is used for device registration. The sponsor has decided not to make it public.